CLINICAL TRIAL: NCT06497686
Title: The Application of Rapid Fresh Digital Pathology on the Diagnosis and Biomarker Testing of Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202405132RINE
Record Dates: First submitted 2024-06-20; First posted 2024-07-12 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Intraoperative Pathology; 3D Pathology; Immunochemistry Staining
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control human lung tissues (normal human lung tissues)
  Interventions: Diagnostic Test: mesoscale nonlinear optical gigascope; Diagnostic Test: Fluorescence microscope
- Cancerous human lung tissues
  Interventions: Diagnostic Test: mesoscale nonlinear optical gigascope; Diagnostic Test: Fluorescence microscope

INTERVENTIONS:
Diagnostic Test: mesoscale nonlinear optical gigascope — An nonlinear optical microscope with ultra-large field of view and ultra-high resolution.
Diagnostic Test: Fluorescence microscope — An optical microscope used to examine the fluorescence signal from stained tissues.

SUMMARY:
Through this project, the rapid staining process will be optimized for ex-vivo human lung specimens and integrate advanced ex-vivo mesoscale nonlinear optical gigascope. Initially, this will provide rapid digital pathological diagnosis during lung cancer surgeries. This will help achieve the dual goals of precise and efficient complete resection of lung cancer tissues while preserving tissue functionality. The application of this technology aims to provide higher-quality medical services for patients suffered from lung cancers.

DETAILED DESCRIPTION:
Frozen section can provide rapid diagnosis during the operation, and its information is very important for surgeons to make decisions for the operative methods, especially for patients whose clinical conditions or lesions sites are inappropriate for biopsy. The frozen section procedure requires a pathological laboratory, a skilled technician, and an experienced pathologist. Not all pathological laboratories can perform the frozen section procedure. The frozen section can also cause frozen artifacts and tissue loss especially for small biopsy samples. In this study rapid fresh digital pathology combining the rapid whole-mount hematoxylin-eosin (H&E) tissue staining (the-RTS) method and optical imaging via mesoscale nonlinear optical gigascope (mNLOG) will be used to obtain digital images with ultra-high resolution of resected lung specimens. These images will be analyzed by experienced pathologists and compared with H&E-stained slides from traditional frozen section procedures to see if the rapid fresh digital pathology can be used as an alternative method for intraoperative frozen section procedure.

Moreover, the potential to use rapid fresh digital pathology in the detection of lung cancer biomarkers (including low-grade or high-grade patterns, invasive or in situ lesions, and STAS) and three-dimensional pathology will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* (1) Adults aged 20 and above.
* (2) Patients diagnosed with lung cancer or lung tumors, scheduled for surgical resection.

A total of 300 patients are expected to be included.

Exclusion Criteria:

* (1) Patients unable to provide consent. (e.g., inability to speak, inability to communicate in Chinese, etc.).
* (2) Patients for whom a definitive pathological diagnosis cannot be established.
* (3) Patients suitable only for biopsy and not for surgical resection.
* (4) Exclude specimens that are too small or lesions that are too small to retain extra tissue.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Following standard surgical procedures for lung cancer tumor resection, the investigators will directly obtain tissue from the post-operative specimens. Without affecting pathological diagnosis, staging, or the assessment of surgical safety margins, the investigators will collect tissue samples measuring approximately 0.5-2.0 cm x 0.5-2.0 cm x 0.3-2.0 cm from the lung cancer/tumor and the surrounding normal tissue or the junction between the tumor and its surrounding normal tissue. These samples will be used for microscopic imaging system detection of lung cancer/tumor tissue. This process, being different from the tissue sent for intraoperative pathological examination, will not affect subsequent diagnosis and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of replacing frozen section pathology with rapid digital pathology diagnosis. | 1 years
  Obtain a portion of specimens and directly perform rapid H&E staining. Then, place the edge of the cut surface of the specimen flat on the microscope objective for observation. The same specimen will then undergo the standard histological staining process in the pathology department for comparative analysis. Another portion of the specimen will be processed using the pathology department's standard frozen section procedure for comparative analysis. In this study, the investigators will acquire the pathological tissue images (with multiple distinct structures like nuclear atypia, vessels, vesicles, and so on) in those images via rapid-fresh-pathology, frozen pathology and formalin-fixed embedded pathology. And the analysis of the number of abnormal cells, irregular vesicles and tumor structures will be conducted to provide pathologists information to compare and distinguish whether it is normal or not.

SECONDARY OUTCOMES:
Utilize rapid digital pathology for biomarker detection and 3D pathology in lung cancer. | 1 year
  Obtain specimens for testing with rapid immunohistochemical (IHC) staining process and used for the three-dimensional reconstruction of lung tissue structure. First, label and stain the specimen using antibodies, then observe it under the mesoscale optical microscope or the fluorescence microscope. The same specimen will then undergo the standard histological staining process in the pathology department for comparative analysis. In this study, the image data will be reconstructed using 3D reconstruction technology to present the three-dimensional structure (for example: vessels, vesicles and so on) of the lung tissue specimen. This will be used for three-dimensional digital pathology research on tumor grading and growth patterns.(including low-grade or high-grade patterns, invasive or in situ lesions, and STAS) and three-dimensional pathology will also be evaluated.

IPD SHARING:
Plan to Share IPD: No